CLINICAL TRIAL: NCT00214630
Title: A 12-week Randomized, Open-label 3-arm, Parallel Group, Multicenter Phase IIIb Study Comparing Efficacy and Safety of Rosuvastatin 20mg and 40mg With That of Atorvastatin 80 mg in Subjects With Acute Coronary Syndromes
Brief Title: LUNAR IIIb Study Comparing Rosuvastatin and Atorvastatin in Subjects With Acute Coronary Syndromes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4522US/0001; D3560L00021; LUNAR
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium; Atorvastatin

INTERVENTIONS:
Drug: rosuvastatin calcium
  Other Names: Crestor
Drug: atorvastatin
  Other Names: Lipitor

SUMMARY:
Comparison of rosuvastatin and atorvastatin in subjects with acute coronary syndromes

ELIGIBILITY:
Inclusion Criteria:

* Non-ST segment elevation ACS and ST segment elevation ACS who receive optimal reperfusion therapy

Exclusion Criteria:

* Previous Q-wave infarct within the last 4 weeks
* CK elevation not caused by myocardial injury
* uncontrolled hypertension at time of randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2003-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Reduction of LDL-C following 12 weeks of treatment

SECONDARY OUTCOMES:
% change from baseline in LDL-C following 2 & 6 weeks of treatment; % change from baseline in TC, HDL-C, triglycerides, non-HDL-C, apolipoprotein A-1, apolipoprotein B, LDL-C/HDL-C, TC/HDL-C, non-HDL-C/HDL-C, ApoB/Apo A-1 @ weeks 6 & 12

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Crestor Medical Science Director, MD, Study Director — AstraZeneca
Locations (56):
- United States (52):
  - Research Site, San Diego, California
  - Research Site, Torrance, California
  - Research Site, Bridgeport, Connecticut
  - Research Site, Atlantis, Florida
  - Research Site, Brandon, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Safety Harbor, Florida
  - Research Site, Tampa, Florida
  - Research Site, Aurora, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Lombard, Illinois
  - Research Site, Melrose Park, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Covington, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Tupelo, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Kalispell, Montana
  - Research Site, Newark, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Rochester, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Fairview Park, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Danville, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Dallas, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Chesapeake, Virginia
  - Research Site, Burien, Washington
  - Research Site, Wausau, Wisconsin
- Research Site, San José, Costa Rica
- Research Site, San Salvador, El Salvador
- Research Site, Ayer, Morocco
- Research Site, Panama City, Panama

REFERENCES:
- [Derived] Pitt B, Loscalzo J, Ycas J, Raichlen JS. Lipid levels after acute coronary syndromes. J Am Coll Cardiol. 2008 Apr 15;51(15):1440-5. doi: 10.1016/j.jacc.2007.11.075. PMID 18402897